CLINICAL TRIAL: NCT02779023
Title: Integrative Cardiac Health Project Cognitive-Behavior Therapy for Insomnia
Acronym: CBT-I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Methodology of subject enrollment would require significant modification.
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 404030
Record Dates: First submitted 2016-04-18; First posted 2016-05-20 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Insomnia; Cardiovascular Risk Factor
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICHP + CBT-I (Experimental): Participants in this arm will receive the usual care (ICHP program) plus 6 Cognitive-Behavior Therapy for Insomnia (CBT-I) treatment sessions. Four of the treatment sessions will be in person and two will be over the phone.
  Interventions: Behavioral: Cognitive-Behavior Therapy for Insomnia (CBT-I)
- ICHP Only (No Intervention): Participants in this arm will receive the usual care (ICHP program).

INTERVENTIONS:
Behavioral: Cognitive-Behavior Therapy for Insomnia (CBT-I)
  Arms: ICHP + CBT-I

SUMMARY:
This study investigates the feasibility, acceptability, and effectiveness of adding Cognitive-Behavioral Therapy for Insomnia (CBT-I) to the standard care received at the Integrative Cardiac Health Project (ICHP) on insomnia symptoms and severity. ICHP is an established cardiovascular disease prevention program to reduce cardiovascular disease risk through the adoption of lifestyle changes related to improvements in diet, stress, sleep, and exercise. The study will be conducted among patients with insomnia who are already enrolled in the ICHP cardiovascular risk prevention program.

This is a single-center study, prospective, randomized, controlled, interventional trial within ICHP at the Walter Reed National Military Medical Center (WRNMMC). To conduct both phases of the study, up to 76 total male and female patients enrolled in ICHP who meet criteria for insomnia will be recruited. Participants who meet inclusion and exclusion criteria for this study, and consent to participate, will be randomized to one of two conditions: (1) ICHP, or (2) ICHP + CBT-I treatment. CBT-I treatment will consist of four in-person appointments and two telephone appointments.

DETAILED DESCRIPTION:
Methodology: Up to 76 total male and female patients enrolled in the ICHP who meet criteria for insomnia will be recruited. All ICHP patients meet the following criteria before enrolling in the program: military beneficiaries at least 18 years of age who are self-referred or referred by their physician.

Randomization: Participants will be selected for treatment groups based on a block randomization scheme. The total number of blocks will be 19, and the number of subjects per block will be 4. The treatment labels will be: ICHP and ICHP + CBT-I. The randomization scheme varies the sequence of treatment categories in each block.

Allocation concealment: The allocation sequence will be concealed from the research team enrolling participants in sequentially numbered, opaque, sealed, and stapled envelopes.

Once randomized, patients identified for the study will participate in the ICHP group or the ICHP + CBT-I group (which consists of the ICHP program plus a 6-session CBT-I treatment). The 6 sessions will consist of 4 in-person appointments and two telephone appointments. Each in-person session will be approximately 1 hour, and each phone session will be approximately 30 minutes.

The study data will be analyzed in two phases. Phase I will be a pilot study to determine the feasibility and acceptability of CBT-I within the ICHP program.

Phase II will be implementation of the full RCT to determine the effectiveness of the CBT-I intervention compared to ICHP usual care. Data collected during Phase I will be utilized in the final analysis unless changes to the procedures which could affect outcome measures are made after participants begin.

Phase I (feasibility and acceptability): Primary outcomes for Phase I of the study will be descriptive statistics on feasibility and acceptability measures as well as qualitative responses to a post-treatment interview with participants. Secondary outcomes for Phase I will be between-group differences in sleep outcomes.

Minimum criteria for advancing to Phase II include the following:

* Recruitment rate: Average of 21 participants enrolled per year. If the recruitment rate during Phase I is not sufficient to enroll 21 participants per year during Phase II, it will be necessary to modify the recruitment strategy in order to increase the rate of participant enrollment before proceeding to Phase II.
* Treatment acceptability rate, as measured by both of the following:

  * 50% of Phase I participants scoring question 3 of the Insomnia Treatment Evaluation Measure-Revised (ITEM-R) as a "3" or "4."
  * Question 3 asks: "How satisfied are you with the treatment received"
  * Minimum of 50% of participants answering question 1 of the Post-Study Questionnaire ("Did you find this insomnia treatment valuable and useful to you?") as: ◦"Yes" (item a) or ◦"Moderately Useful" (item c)

Phase II (effectiveness of intervention): Primary outcomes for Phase II will be between-group differences in level of change in sleep outcomes. Secondary outcomes for Phase II will include: between-group differences in changes in depression, fatigue, perceived stress, sleepiness, and sleep-related quality of life. Tertiary outcomes (exploratory) will include changes in secondary cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older, Tricare beneficiary, participation in ICHP
* Sleep-onset or maintenance insomnia, defined as sleep-onset latency (SOL; time it takes to fall asleep) and/or wake after sleep onset (WASO; time spent awake after falling asleep) longer than 30 minutes per night at least 3 nights per week
* Insomnia duration of at least 3 months
* A complaint of at least 1 negative effect during waking hours (e.g., fatigue, impaired functioning, mood disturbances) that is attributed to insomnia
* Score of 8 or greater on the Insomnia Severity Index
* Pittsburgh Sleep Quality Index (PSQI) score of > 5

Exclusion Criteria:

* Previous participation in the ICHP program
* Use of stimulant medications or acute high dose of steroids
* Suicidal ideation, as determined by a score of 1 or greater on question #9 of the Patient Health Questionnaire-9 (PHQ-9)
* Concurrent psychological or behavioral treatment for insomnia
* Current pregnancy by history, or plans to become pregnant in the next 6 months (excluded because of sleep difficulties which often occur during pregnancy that could confound the results)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | 2 months, 4 months, and 6 months
  collected through sleep diary and actigraphy

SECONDARY OUTCOMES:
Insomnia Severity Index | 2 months, 4 months, and 6 months
  7-item self report measure of insomnia symptoms
Perceived Stress | 2 months, 4 months, and 6 months
  14-item self report of perceived stress
Patient Health Questionnaire-9 | 2 months, 4 months, and 6 months
  9-item self report measure of depressive symptoms
Multidimensional Fatigue Inventory | 2 months, 4 months, and 6 months
  20-item self report measure of fatigue
Epworth Sleepiness Scale | 2 months, 4 months, and 6 months
  7-item self report measure of sleepiness
Functional Outcomes of Sleep Questionnaire-10 | 2 months and 6 months
  10-item self report measure of the effect of sleepiness on daytime function
Pittsburgh Sleep Quality Index | 2 months and 6 months
  11-item self report measure of sleep quality

OTHER OUTCOMES:
Insomnia Treatment Acceptability Scale-Behavior Subscale | 2 weeks and again at 2 months
  8-item self report measure of perceived treatment acceptability
Insomnia Treatment Evaluation Measure-Revised | 2 months
  6-item self report measure of the credibility and effectiveness of the insomnia treatment

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Villines, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Integrative Cardiac Health Project, Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No